CLINICAL TRIAL: NCT07124130
Title: Parenteral Lactated Ringer's Plus Dextrose 5% vs Lactated Ringer's in Labor: A Randomized Control Trial on Maternal and Neonatal Outcomes
Brief Title: Lactated Ringer's and Dextrose 5% vs Only Lactated Ringer's in Labor
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Tetsuya Kawakita, MD, Associate Professor, Eastern Virginia Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-03-FB-0052
Record Dates: First submitted 2025-07-22; First posted 2025-08-15 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Induced Labor
Keywords: Induced labor; 5% dextrose; Lactated Ringers; duration of labor
MeSH Terms: interventions — Glucose; Ringer's Lactate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 5% dextrose and Lactate Ringer (Active Comparator): Participants randomized to this arm will receive an intravenous solution of 5% dextrose and Lactate Ringer during labor.
  Interventions: Drug: 5% Dextrose (D5) in Normal Saline (NS); Drug: Lactate Ringer
- Lactate Ringer only (Active Comparator): Participants randomized to this arm will receive an intravenous Lactate Ringer solution only.
  Interventions: Drug: Lactate Ringer

INTERVENTIONS:
Drug: 5% Dextrose (D5) in Normal Saline (NS) — A solution of 5% dextrose and lactate ringer will be given to one group of participants.
  Arms: 5% dextrose and Lactate Ringer
Drug: Lactate Ringer — A Lactate Ringer solution will be given to one group of participants.

SUMMARY:
The goal of this clinical trial is to determine which of two types of standard intravenous (IV) fluids (a combination of 5% dextrose and Lactated Ringers solution and Lactated Ringers solution alone) has a better influence on labor when inducing labor in pregnant women. The main questions it aims to answer are:

1. Does the use of 5% dextrose and Lactated Ringers lead to a shorter labor than the use of just Lactated Ringers?
2. Does the use of 5% dextrose and Lactated Ringers increase the risk of neonatal hypoglycemia when compared to Lactated Ringers? Participants in this trial will be randomly assigned to one of two groups: a group that receives a solution of 5% dextrose and Lactated Ringers, and a group that receives Lactated Ringers alone. Researchers will compare the outcomes of the two groups to see which IV fluid is more effective.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women
* Age 18 years or older and able to provide informed consent
* Singleton pregnancy at term
* Induction of labor
* Cephalic presentation
* Unfavorable cervix (Bishop score ≤ 6)

Exclusion Criteria:

* Age under 18 years
* Involuntarily confined or detained
* Considered as having diminished decision-making capacity
* Spontaneous labor (cervical exam between 5-6 cm) with or without ruptured membraned
* Favorable cervix (Bishop score >6)
* Diabetes mellitus (both gestational and pre-gestational)
* Structural renal disease
* Acute or chronic kidney disease resulting in abnormal creatinine or proteinuria
* Evidence of chorioamnionitis or non-reassuring fetal testing at the time of enrollment
* Pyrexia (>38.0 degrees Celsius)
* Stillbirth
* Planned cesarean delivery
* Women presenting with emergent circumstances for labor induction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Time from Induction Start To Delivery | From enrollment to the end of labor

SECONDARY OUTCOMES:
Type of amniotomy | From enrollment until delivery
  Spontaneous vs artificial
Mode of Delivery | From enrollment until delivery.
  The incidence of spontaneous vaginal delivery, operative vaginal delivery and cesarean delivery.
Indication for cesarean delivery | From enrollment until delivery.
  Rate of failed induction of labor, arrest of active phase, arrest of descent, non-reassuring fetal condition, maternal request, other.
Delivery within 12 hours of induction. | Time from induction until delivery.
  Incidence of delivery within 12 hours of induction.
Delivery within 24 hours of Induction | Time of induction to time of delivery.
  Incidence of delivery within 24 hours of induction.
Delivery within 36 hours of Induction | From time of induction to time of delivery.
  Incidence of delivery within 36 hours of induction.
Delivery within 48 hours of Induction | From time of induction to time of delivery.
  Incidence of delivery within 48 hours of induction.
Perineal Lacerations (Degree I-IV) | From time of enrollment to time of delivery.
  Degree of perineal lacerations occurring during delivery (first to fourth degree).
Postpartum hemorrhage | Time of enrollment to time of delivery.
  Blood loss >1000 mL
Blood Transfusion | From time of enrollment to hospital discharge (up to 42 days post-delivery).
  Incidence of blood transfusions required during or after delivery.
Isolated maternal fever | From time of enrollment to hospital discharge (up to 42 days post-delivery).
  Incidence of maternal fever (T>38°C)
Diagnosed Endometritis | From time of enrollment to hospital discharge (up to 42 days post-delivery).
  The number of endometritis based on clinical signs and diagnostic tests.
Wound Separation/Infection | From time of enrollment to hospital discharge (up to 42 days post-delivery).
  Incidence of wound separation or infection requiring additional closure or antibiotics.
Intraamniotic Infection | From time of enrollment to hospital discharge (up to 42 days post-delivery).
  Presence of maternal fever, tachycardia, and/or fundal tenderness suggesting intraamniotic infection.
Venous Thromboembolism (VTE) | From time of enrollment to hospital discharge (up to 42 days post-delivery).
  Occurrence of venous thromboembolism.
Hysterectomy | From time of enrollment to hospital discharge (up to 42 days post-delivery).
  Occurrence of hysterectomy related to delivery complications.
Intensive Care Unit (ICU) Admission | From time of enrollment to ICU admission (up to 42 days post-delivery).
  Admission to ICU for maternal complications.
Maternal Death | From time of enrollment until maternal death (up to 42 days post-delivery).
  Occurrence of maternal death during or after delivery.
Length of hospital stay | From time of hospital admission to time of hospital discharge (up to 50 days post-delivery).
  Days between admission and discharge
Cord Prolapse | From time of enrollment to delivery.
  Occurrence of cord prolapse during labor.
Use of Terbutaline | From time of enrollment to delivery.
  The number of terbutaline use for uterine contractions.
Placement of Intrauterine Pressure Catheter | From time of enrollment to delivery.
  The number of placement of intrauterine pressure catheter during labor.
Epidural Use | From time of enrollment to delivery.
  Use of epidural anesthesia during labor for pain relief.
Neonatal Severe Respiratory Distress Syndrome (RDS) | From time of delivery to hospital discharge. Includes the entire length of neonate's hospital stay, up to 1 year following delivery.
  Need for intubation and mechanical ventilation for ≥12 hours.
Neonatal 5- minute Apgar score <7 | From time of delivery up to 1 day following delivery.
  Incidence of 5-minute Apgar score<7
Arterial umbilical cord pH <7 | From time of enrollment up to 1 day following delivery.
  Incidence of arterial umbilical cord pH <7
Neonatal outcome composite | From time of delivery to hospital discharge. Includes the entire length of neonate's hospital stay, up to 1 year following delivery.
  Incidence of neonatal outcome composite
Neonatal Sepsis (Culture-proven or Presumed) | From time of delivery to hospital discharge. Includes the entire length of neonate's hospital stay, up to 1 year following delivery.
  Incidence of neonatal sepsis, culture-proven or presumed.
Neonatal Intensive Care Unit (NICU) Admission | From time of delivery to NICU admission. Includes the entire length of neonate's hospital stay, up to 1 year following delivery.
  Admission of neonate to NICU.
Hypoxic-Ischemic Encephalopathy | From time of delivery to hospital discharge. Includes the entire length of neonate's hospital stay, up to 1 year following delivery.
  Diagnosis of hypoxic-ischemic encephalopathy in neonates.
Neonatal Intraventricular Hemorrhage (Grade 3 or 4) | From time of enrollment to hospital discharge. Includes the entire length of neonate's hospital stay, up to 1 year following delivery.
  Occurrence of grade 3 or 4 intraventricular hemorrhage in neonates.
Diagnosed Neonatal Necrotizing Enterocolitis | From time of delivery to time of hospital discharge. Includes the entire length of neonate's hospital stay, up to 1 year following delivery.
  The number of diagnosis of necrotizing enterocolitis in the neonate.
Neonatal Head Cooling Therapy | From time of delivery to time of hospital discharge. Includes the entire length of neonate's hospital stay, up to 1 year following delivery.
  Use of head cooling therapy for neonates to prevent brain injury.
Neonatal Blood Transfusion | From time of delivery to time of hospital discharge. Includes the entire length of neonate's hospital stay, up to 1 year following delivery.
  Need for blood transfusion in the neonate.
NICU Stay >48 hours | From NICU admission to NICU discharge. Includes the entire length of neonate's hospital stay, up to 1 year following delivery.
  Incidence of NICU stay lasting longer than 48 hours.
Neonatal Length of Stay (days) | From time of delivery to time of hospital discharge. Includes the entire length of neonate's hospital stay, up to 1 year following delivery.
  Total length of neonatal stay in the hospital.
Bishop Score: Cervical Dilation, Effacement, Station, Position, Consistency | From time of enrollment to time of induction up to 1 week.
  Baseline Bishop score (0-13, with 13 being more favorable to labor) and its changes during labor to assess cervical readiness for induction.

CONTACTS AND LOCATIONS:
Locations (2):
- Sentara Norfolk General Hospital, Norfolk, Virginia, United States
- Policlinico di Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greenland S. Avoiding power loss associated with categorization and ordinal scores in dose-response and trend analysis. Epidemiology. 1995 Jul;6(4):450-4. doi: 10.1097/00001648-199507000-00025. No abstract available. PMID 7548361
- [Background] Carbone JF, Tuuli MG, Fogertey PJ, Roehl KA, Macones GA. Combination of Foley bulb and vaginal misoprostol compared with vaginal misoprostol alone for cervical ripening and labor induction: a randomized controlled trial. Obstet Gynecol. 2013 Feb;121(2 Pt 1):247-252. doi: 10.1097/AOG.0b013e31827e5dca. PMID 23303106
- [Background] Moraes Filho OB, Albuquerque RM, Cecatti JG. A randomized controlled trial comparing vaginal misoprostol versus Foley catheter plus oxytocin for labor induction. Acta Obstet Gynecol Scand. 2010 Aug;89(8):1045-52. doi: 10.3109/00016349.2010.499447. PMID 20636243
- [Background] Gomez Slagle HB, Fonge YN, Caplan R, Pfeuti CK, Sciscione AC, Hoffman MK. Early vs expectant artificial rupture of membranes following Foley catheter ripening: a randomized controlled trial. Am J Obstet Gynecol. 2022 May;226(5):724.e1-724.e9. doi: 10.1016/j.ajog.2021.11.1368. Epub 2022 Feb 6. PMID 35135684
- [Background] Berry M, Lamiman K, Slan MN, Zhang X, Arena Goncharov DD, Hwang YP, Rogers JA, Pacheco LD, Saade GR, Saad AF. Early vs delayed amniotomy following transcervical Foley balloon in the induction of labor: a randomized clinical trial. Am J Obstet Gynecol. 2024 May;230(5):567.e1-567.e11. doi: 10.1016/j.ajog.2024.01.028. Epub 2024 Feb 15. PMID 38367749
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509
- [Background] WHO recommendations: Intrapartum care for a positive childbirth experience. Geneva: World Health Organization; 2018. Available from http://www.ncbi.nlm.nih.gov/books/NBK513809/ PMID 30070803
- [Background] Shafaie FS, Mohaddesi H, Mirghafourvand M, Yulghunlu FA. A randomized, double-blinded, controlled trial comparing parenteral dextrose 5%, Ringer's solution and oral intake on the delivery outcomes in nulliparas. Int J Womens Health 2017;283-9.
- [Background] Cowett RM, Susa JB, Giletti B, Oh W, Schwartz R. Glucose kinetics in infants of diabetic mothers. Am J Obstet Gynecol. 1983 Aug 1;146(7):781-6. doi: 10.1016/0002-9378(83)91077-3. PMID 6346883
- [Background] Dapuzzo-Argiriou LM, Smulian JC, Rochon ML, Galdi L, Kissling JM, Schnatz PF, Gonzalez Rios A, Airoldi J, Carrillo MA, Maines J, Kunselman AR, Repke J, Legro RS. A multi-center randomized trial of two different intravenous fluids during labor. J Matern Fetal Neonatal Med. 2016;29(2):191-6. doi: 10.3109/14767058.2014.998190. Epub 2015 Sep 4. PMID 25758624
- [Background] Cerri V, Tarantini M, Zuliani G, Schena V, Redaelli C, Nicolini U. Intravenous glucose infusion in labor does not affect maternal and fetal acid-base balance. J Matern Fetal Med. 2000 Jul-Aug;9(4):204-8. doi: 10.1002/1520-6661(200007/08)9:43.0.CO;2-9. PMID 11048829
- [Background] Fisher AJ, Huddleston JF. Intrapartum maternal glucose infusion reduces umbilical cord acidemia. Am J Obstet Gynecol. 1997 Oct;177(4):765-9. doi: 10.1016/s0002-9378(97)70265-5. PMID 9369816
- [Background] Pare J, Pasquier JC, Lewin A, Fraser W, Bureau YA. Reduction of total labor length through the addition of parenteral dextrose solution in induction of labor in nulliparous: results of DEXTRONS prospective randomized controlled trial. Am J Obstet Gynecol. 2017 May;216(5):508.e1-508.e7. doi: 10.1016/j.ajog.2017.01.010. Epub 2017 Jan 30. PMID 28153654
- [Background] Philipson EH, Kalhan SC, Riha MM, Pimentel R. Effects of maternal glucose infusion on fetal acid-base status in human pregnancy. Am J Obstet Gynecol. 1987 Oct;157(4 Pt 1):866-73. doi: 10.1016/s0002-9378(87)80075-3. PMID 3314516
- [Background] Collinot H, Merrer J, Girault A, Goffinet F, Le Ray C. Implementation of glucose 5% supplementation protocol to reduce the duration of labor among women with cervical ripening by prostaglandins: The GLUCOSHORT before-and-after study. J Gynecol Obstet Hum Reprod. 2023 May;52(5):102558. doi: 10.1016/j.jogoh.2023.102558. Epub 2023 Feb 19. PMID 36806716
- [Background] Sharma C, Kalra J, Bagga R, Kumar P. A randomized controlled trial comparing parenteral normal saline with and without 5% dextrose on the course of labor in nulliparous women. Arch Gynecol Obstet. 2012 Dec;286(6):1425-30. doi: 10.1007/s00404-012-2485-1. Epub 2012 Aug 4. PMID 22865033
- [Background] Shrivastava VK, Garite TJ, Jenkins SM, Saul L, Rumney P, Preslicka C, Chan K. A randomized, double-blinded, controlled trial comparing parenteral normal saline with and without dextrose on the course of labor in nulliparas. Am J Obstet Gynecol. 2009 Apr;200(4):379.e1-6. doi: 10.1016/j.ajog.2008.11.030. Epub 2009 Feb 14. PMID 19217592
- [Background] Hernandez Lopez AB, Muriel Miguel C, Fernandez-Canadas Morillo A, Lopez Lapeyrere C, Perez Medina T, Salcedo Marina A, Fornet Ruiz I, Rubio Gonzalez E, Solis Munoz M. Efficacy of "optimal hydration" during labor: HYDRATA study protocol for a randomized clinical trial. Res Nurs Health. 2020 Jan;43(1):8-16. doi: 10.1002/nur.21998. Epub 2019 Dec 2. PMID 31793019
- [Background] Nordstrom L, Arulkumaran S, Chua S, Ratnam S, Ingemarsson I, Kublickas M, Persson B, Shimojo N, Westgren M. Continuous maternal glucose infusion during labor: effects on maternal and fetal glucose and lactate levels. Am J Perinatol. 1995 Sep;12(5):357-62. doi: 10.1055/s-2007-994496. PMID 8540943
- [Background] Riegel M, Quist-Nelson J, Saccone G, Locci M, Shrivastava VK, Salim R, Fisher A, Nordstrom L, Kunselman AR, Repke J, Fong A, Smulian J, Xodo S, Mokhtari N, Zullo F, Berghella V. Dextrose intravenous fluid therapy in labor reduces the length of the first stage of labor. Eur J Obstet Gynecol Reprod Biol. 2018 Sep;228:284-294. doi: 10.1016/j.ejogrb.2018.07.019. Epub 2018 Jul 17. PMID 30055509
- [Background] Stratton JF, Stronge J, Boylan PC. Hyponatraemia and non-electrolyte solutions in labouring primigravida. Eur J Obstet Gynecol Reprod Biol. 1995 Apr;59(2):149-51. doi: 10.1016/0028-2243(95)02042-q. PMID 7657008
- [Background] Oral E, Gezer A, Cagdas A, Pakkal N. Oxytocin infusion in labor: the effect different indications and the use of different diluents on neonatal bilirubin levels. Arch Gynecol Obstet. 2003 Jan;267(3):117-20. doi: 10.1007/s00404-002-0298-3. PMID 12552319
- [Background] Omigbodun AO, Akindele JA, Osotimehin BO, Fatinikun T, Fajimi JL, Adeleye JA. Effect of saline and glucose infusions of oxytocin on neonatal bilirubin levels. Int J Gynaecol Obstet. 1993 Mar;40(3):235-9. doi: 10.1016/0020-7292(93)90836-l. PMID 8096475
- [Background] Garmi G, Zuarez-Easton S, Zafran N, Ohel I, Berkovich I, Salim R. The effect of type and volume of fluid hydration on labor duration of nulliparous women: a randomized controlled trial. Arch Gynecol Obstet. 2017 Jun;295(6):1407-1412. doi: 10.1007/s00404-017-4381-1. Epub 2017 May 3. PMID 28470550
- [Background] Loong EP, Lao TT, Chin RK. Effects of intrapartum intravenous infusion of 5% dextrose or Hartmann's solution on maternal and cord blood glucose. Acta Obstet Gynecol Scand. 1987;66(3):241-3. doi: 10.3109/00016348709020755. PMID 3310504
- [Background] Fong A, Serra AE, Caballero D, Garite TJ, Shrivastava VK. A randomized, double-blinded, controlled trial of the effects of fluid rate and/or presence of dextrose in intravenous fluids on the labor course of nulliparas. Am J Obstet Gynecol. 2017 Aug;217(2):208.e1-208.e7. doi: 10.1016/j.ajog.2017.03.010. Epub 2017 Mar 18. PMID 28322776
- [Background] Ahadi Yulghunlu F, Sehhatie Shafaie F, Mirghafourvand M, Mohaddesi H. The effects of intravenous dextrose 5%, Ringer's solution, and oral intake on the duration of labor stages in nulliparous women: a double-blind, randomized, controlled trial. J Matern Fetal Neonatal Med. 2020 Jan;33(2):289-296. doi: 10.1080/14767058.2018.1489792. Epub 2018 Sep 9. PMID 29909704

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT07124130/Prot_SAP_000.pdf
  • Informed Consent Form (2025-05-19): https://cdn.clinicaltrials.gov/large-docs/30/NCT07124130/ICF_001.pdf